CLINICAL TRIAL: NCT06307275
Title: The Effect of Intermittent Fasting on Body Fat and Quality of Life
Brief Title: Intermittent Fasting on Body Fat and Quality of Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 5170221
Record Dates: First submitted 2024-02-29; First posted 2024-03-12 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non Fasting (Active Comparator): For four week: Participants will keep their normal food intake with no restrictions on when to eat. Participants will keep their normal weekly exercise routine.
  Interventions: Other: non fasting
- Fasting (Experimental): For four weeks: Fasting for 16 hours from participant last meal of the previous evening's meal to the first meal of the next day. Then for 8 hours, participant is able to eat. During the fasting, participants are allowed to consume water and black coffee/tea. Participants will also keep their normal weekly exercise routine.
  Interventions: Other: Fasting

INTERVENTIONS:
Other: Fasting — Fasting for 16 hours from participant last meal of the previous evening's meal to the first meal of the next day. Then for 8 hours, participant is able to eat. During the fasting, participants are allowed to consume water and black coffee/tea. Participants will also keep their normal weekly exercise routine.
  Arms: Fasting
Other: non fasting — Participants will not be fasting during these four weeks. They will eat their normal food intake and keep their normal physical activity levels.
  Arms: Non Fasting

SUMMARY:
The purpose of this investigator-initiated study to check the feasibility that intermittent fasting has on body fat loss and quality of life.

DETAILED DESCRIPTION:
Start of study: Informed Consent, Body Fat Analysis, Questionnaires on quality of life, sleep, and stress. For the next four weeks, participants will eat their normal food intake with no restrictions on when to eat. Participants will keep their normal weekly exercise routine.

Midway of study: Body Fat Analysis, Questionnaires on quality of life, sleep, and stress. For the next four weeks, participants will do the intermittent fasting program. This program has participants fasting 16 hours from their last meal of the previous evening's meal to the first meal of their next day. Then for 8 hours, participants are able to eat. During the fasting, participants are allowed to consume water and black coffee/tea. Participants will also keep their normal weekly exercise routine.

End of study: Body Fat Analysis, Questionnaires on quality of life, sleep, and stress.

ELIGIBILITY:
Inclusion Criteria:

• In good health

Exclusion Criteria:

• Diabetes or Metabolic Syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Body fat percentage | change between baseline and eight weeks
  Body composition will give the following measurement: body fat percentage
Visceral fat | change between baseline and eight weeks
  In addition, body composition will also give us visceral fat measurement

CONTACTS AND LOCATIONS:
Overall Officials: Gurinder Bains, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States